CLINICAL TRIAL: NCT01270555
Title: Efficacy Of Bupropion SR For Attention Deficit Hyperactivity Disorder (ADHD) In Adults With Recent Past or Current Substance Use Disorders
Brief Title: Efficacy Of Bupropion For Attention Deficit Hyperactivity Disorder (ADHD) In Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Timothy Wilens, MD, MD, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1999-P-009198; NCT01012024 (obsolete NCT alias)
Record Dates: First submitted 2011-01-03; First posted 2011-01-05 (Estimated); Results first posted 2011-02-25 (Estimated); Last update posted 2013-03-08 (Estimated); Status verified 2013-03

CONDITIONS: Attention Deficit Hyperactivity Disorder (ADHD); Substance Use Disorder (SUD)
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity; Substance-Related Disorders | interventions — Bupropion

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Bupropion (Experimental)
  Interventions: Drug: Bupropion SR

INTERVENTIONS:
Drug: Bupropion SR — 100mg capsules Initial dosing 100mgSR every morning, to be titrated to 200mgSR twice daily maximum
  Other Names: Wellbutrin

SUMMARY:
The investigators propose to conduct an open study to evaluate the efficacy and tolerability of Bupropion SR using clinically relevant doses in ADHD adults with a recent history of or current substance use disorders. We hypothesize that Bupropion SR will be effective in treating ADHD in this population.

ELIGIBILITY:
Inclusion Criteria:

* Male and female outpatients 18 years old or older, up to 60 years old.
* Patients with the diagnosis of Attention Deficit Hyperactivity Disorder (ADHD), by DSM-IV, as manifested in clinical evaluation and confirmed by structured interview.
* Patients within the past 6 months known to abuse or to be dependent on alcohol or any drug (nicotine addiction not included)

Exclusion Criteria:

* Any clinically unstable medical condition
* Clinically significant abnormal baseline laboratory values
* Mental retardation (I.Q. <75) or Organic brain disorders
* Seizure disorder
* Patients with a history or an eating disorder including anorexia or bulimia nervosa
* Pregnant or nursing females
* Patients with current bipolar disorder
* Psychotic disorder of any type
* Patients on psychotropics known to treat ADHD (i.e. stimulants, tricyclics)
* Patients receiving psychotherapy known to treat ADHD (i.e. cognitive or cognitive/behavioral psychotherapy)
* Patients demonstrating active withdrawal from substance abuse

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 1999-05; Primary Completion 2001-07 (Actual)

RESULTS

PARTICIPANT FLOW:
Groups:
- Bupropion: Once daily treatment with Bupropion with intention to treat ADHD and SUD.
Period: Overall Study
Arm/Group | Bupropion
Started | 32
Completed | 19
Not Completed | 13

BASELINE CHARACTERISTICS:
Arm/Group | Bupropion
Number analyzed (Participants) | 32
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 32
  >=65 years | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 32 (8.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 26
Region of Enrollment [Number; unit: participants]
  United States | 32
DSM-IV Attention Deficit Hyperactivity Rating Scale (ADHD RS) [Mean (Standard Deviation); unit: Units on a scale] — Assesses 18 individual criteria symptoms on a severity grid (0=not present, 3=severe; overall minimum score = 0, maximum score = 54)
  Units on a scale | 34.1 (8.2)
Self-reported Weekly substance use [Number; unit: Participants] — Participants who self-report using at least one of illegal drugs or alcohol, at least once per week.
  Participants | 32
Clinical Global Impressions (CGI) Score for SUD Severity [Mean (Standard Deviation); unit: Units on a scale] — Global Severity 1=not ill, 7=extremely ill
  Units on a scale | 4.0 (0.9)
Clinical Global Impressions (CGI) Score for ADHD Severity [Mean (Standard Deviation); unit: Units on a scale] — Global Severity 1=not ill, 7=extremely ill
  Units on a scale | 5.0 (0.7)
Hamilton Anxiety Rating Scale (HAM-A) [Mean (Standard Deviation); unit: Units on a scale] — minimum (least severe anxiety) = 0, maximum (most severe) = 56
  Units on a scale | 8.1 (6.5)
Hamilton Depression rating Scale (HAM-D) [Mean (Standard Deviation); unit: Units on a scale] — minimum (least severe depression) = 0, maximum (most severe) = 84
  Units on a scale | 8.8 (9.1)
Beck Depression Inventory (BDI) [Mean (Standard Deviation); unit: Units on a scale] — minimum (least severe depression) = 0, maximum (most severe) = 63
  Units on a scale | 8.9 (5.9)

OUTCOME MEASURES:

1. Primary Outcome: Attention Deficit Hyperactivity Disorder Rating Scale (ADHD-RS) Score
Description: Assesses 18 individual criteria symptoms using a severity grid (0 = not present, 3 = severe; overall minimum score = 0, maximum score = 54)
Time Frame: baseline and six weeks
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Bupropion
Number analyzed (Participants) | 32
Units on a scale | 19.4 (11.4)

2. Secondary Outcome: Clinical Global Impressions (CGI) Scale of Substance Use Disorder (SUD) Severity
Description: CGI-S 1=not ill, 7=extremely ill
Time Frame: baseline and six weeks
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Bupropion
Number analyzed (Participants) | 32
Units on a scale | 3.1 (0.8)

3. Secondary Outcome: Clinical Global Impressions (CGI) Scale of ADHD Severity
Description: Global Severity (CGI-S) 1=not ill, 7=extremely ill
Time Frame: baseline and six weeks
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Bupropion
Number analyzed (Participants) | 32
Units on a scale | 3.8 (1.1)

4. Primary Outcome: Self-reported Weekly Substance Use
Description: Number of subjects who self-report using at least one of illegal drugs or alcohol, at least once in a week.
Time Frame: baseline and six weeks
Measure: Number; unit: Participants
Arm/Group | Bupropion
Number analyzed (Participants) | 18
Participants | 18

5. Secondary Outcome: Hamilton Anxiety Scale (HAM-A)
Description: minimum score (least severe anxiety) = 0, maximum (most severe) = 56
Time Frame: baseline and six weeks
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Bupropion
Number analyzed (Participants) | 32
Units on a scale | 4.5 (6.9)

6. Secondary Outcome: Hamilton Depression Scale (HAM-D)
Description: minimum score (least severe depression) = 0, maximum score (most severe) = 84
Time Frame: baseline and six weeks
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Bupropion
Number analyzed (Participants) | 32
Units on a scale | 4.5 (5.7)

7. Secondary Outcome: Beck Depression Inventory (BDI)
Description: minimum score (least severe depression) = 0, maximum score (most severe) = 63
Time Frame: baseline and six weeks
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Bupropion
Number analyzed (Participants) | 32
Units on a scale | 3.7 (5.1)

ADVERSE EVENTS:
Arm/Group | Bupropion
Serious Adverse Events (participants affected / at risk) | 0/32
Other Adverse Events (participants affected / at risk) | 0/32

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No